CLINICAL TRIAL: NCT00702494
Title: An Open, Phase I, Dose Escalation Study of the Monoclonal Antibody TB-403 Directed Against PlGF, Given as Multiple IV-doses to Patients With Solid Tumors.
Brief Title: Phase I Study on Monoclonal Antibody TB-403 Directed Against PlGF in Patients With Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioInvent International AB (Industry)
Collaborators: Oxurion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-TB-403-02; EUDRACT No: 2008-001345-25
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2022-03-16 (Actual); Status verified 2009-12

CONDITIONS: Solid Tumors
Keywords: placental growth factor; monoclonal antibody; Phase I; solid tumors; Patients with solid tumors
MeSH Terms: interventions — TB-403

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Multiple IV doses of TB-403, an antibody directed against PlGF
  Interventions: Biological: TB-403

INTERVENTIONS:
Biological: TB-403 — Multiple IV

SUMMARY:
TB-403 is a monoclonal antibody directed against Placental Growth Factor (PlGF). The antibody binds to PlGF and inhibits the binding to it's receptor, VEGF-1. By preventing this binding, growth of tumor vessels are inhibited and tumor growth prevented.

In this study we are investigating the tolerability and safety of TB-403 in patients with solid tumors who receives multiple intravenous doses of TB-403.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed malignity
* Measurable disease
* Performance status 1 or less (ECOG)

Exclusion Criteria:

* Acute illness or infection
* Concurrent second malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of an anti-PlGF antibody | 85 days

SECONDARY OUTCOMES:
Determine multiple dose IV pharmacokinetics | 85 days

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Lassen, MD, PhD, Study Chair — Rigshospitalet, Denmark; Lena Winstedt, PhD, Study Director — BioInvent International AB; Dorthe Nielsen, MD, PhD, Principal Investigator — Herlev Hospital, Herlev, Denmark
Locations (2):
- Denmark (2):
  - Onkologisk Klinik 5072 Finsencentret Rigshospitalet, Copenhagen
  - Onkologisk Afdeling 54B1 Herlev Hospital, Herlev